CLINICAL TRIAL: NCT00763178
Title: Effects of Duloxetine on Fear Conditioning in PTSD
Brief Title: Effects of Duloxetine on Fear Conditioning in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0612002110; M120627
Record Dates: First submitted 2007-12-25; First posted 2008-09-30 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTSD (Experimental): Duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Dosage given according to the following schedule:
  Week 1: 30mg QD, Week 2: 60mg QD, Week 3: 60mg QD, Week 4-6: Flexible dosing according to clinical situation, dose range between 60-120mg QD, Weeks 7 + 8: fixed dose
  Other Names: Cymbalta

SUMMARY:
Chronic posttraumatic stress disorder (PTSD) is a debilitating disorder and treatment response to pharmacological interventions has been modest for these patients. Chronic elevated anxiety and associated psychophysiological parameters including increased heart rate and alterations in skin conductance are key symptoms of chronic PTSD. Selective serotonin reuptake inhibitors (SRIs) are considered treatment of first choice for these patients, however a substantial portion of patients treated with SRIs do not respond sufficiently. Therefore, there is a need to establish novel and effective treatment strategies for these patients. Recently, duloxetine has received considerable attention since it was shown in multiple controlled trials to be an effective treatment for people with major depressive disorder (MDD), a condition which is often co-morbid with PTSD. In chronic PTSD, the psychophysiological responses at baseline and in response to treatment with duloxetine have been inadequately studied and may provide novel insight into antidepressant and anxiolytic mechanisms of this compound.

Primary Aim 1: Evaluate the anxiolytic and antidepressant effects of duloxetine in patients with chronic PTSD.

Secondary Aim 2: Evaluate the effects of duloxetine on fear conditioned psychophysiological responses (including startle eyeblink, skin conductance, and cardiovascular inter-beat interval) at baseline and after 8 weeks of naturalistic treatment in chronic PTSD patients.

ELIGIBILITY:
Inclusion criteria:

* Patients with PTSD (age range 18-65 years) as determined by the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, non-patient version (First et al., 1996)
* Willingness to participate in a naturalistic treatment study using duloxetine and in two fear conditioning tests, one at baseline and one at the end of the 8 weeks treatment study. We will include PTSD subjects on medications (possible medications include antidepressants, benzodiazepines, and neuroleptics) who have no or only partial treatment response or PTSD patients who are untreated. Treatment will be switched to duloxetine and the previous antidepressant medication will be discontinued.
* PTSD subjects will have a minimum score of 50 on the Clinician-Administered PTSD Scale (CAPS; Blake et al, 1995).
* Participants will be enrolled until the number of 20 subjects who complete the study is reached.
* All subjects are required to be in a medically stable condition as determined by a thorough physical examination, including ECG, blood work and urine analysis.
* No vulnerable subjects will be recruited for this study.

Exclusion criteria:

* comorbid diagnosis of bipolar illness, schizophrenia or other psychotic disorders or presence of psychotic symptoms
* acute or chronic suicidality
* acute or chronic unstable medical conditions (including severely impaired hepatic function as indicated with abnormal PT and PTT, abnormal CBC, and liver enzymes more than 50% above the upper normal range, not well controlled blood pressure)
* current diagnosis of substance abuse or dependence
* unsuccessful treatment history with duloxetine, known hypersensitivity to duloxetine or any of its inactive ingredients
* administration of any investigational drug up to 90 days before entry into the study
* intake of monoamino oxides inhibitors up to 90 days before entry into the study or during the study
* subjects with a positive screen for drugs of abuse
* no startle or skin conductance response, or excessively high startle response to the startle probe (100 dB acoustic stimuli) during the pretest
* patients with uncontrolled narrow-angle glaucoma
* Pregnant as indicated by urine pregnancy test or unwillingness to prevent conception during the course of the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Anxiolytic and antidepressant effects of duloxetine in patients with chronic PTSD | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Neumeister, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States